CLINICAL TRIAL: NCT05036252
Title: A Pilot Study of Cardiopulmonary Exercise Testing in Patients With Left Ventricular Systolic Dysfunction Receiving HER2-Targeted Therapy
Brief Title: Study of Cardiopulmonary Exercise Testing in Women Who Have HER2-Positive Breast Cancer With Mild Cardiotoxicity
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-271
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; HER2-positive Metastatic Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Stage IV; Cardiotoxicity
Keywords: HER2-positive breast cancer; cardiotoxicity; HER2-targeted therapy; Breast cancer; 21-271; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Exercise Test; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Participants with HER2-positive breast cancer: Participants with HER2-positive breast cancer who have developed mild cardiotoxicity during HER2-targeted therapy, defined by a decline in LVEF > 10% to < 53% without symptoms of clinical heart failure (NYHA class III or IV), will be eligible for participation in this study.
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Test; Diagnostic Test: Echocardiogram; Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Test — All enrolled participants will undergo a cardiopulmonary exercise test (CPET). The CPET will be conducted using an electronic motorized treadmill with 12-lead ECG monitoring performed by ACSM-certified exercise physiologists.
  Other Names: CPET
Diagnostic Test: Echocardiogram — Resting assessment of LVEF and GLS will be evaluated through Conventional 2D and Doppler echocardiograms will be performed per protocol using a commercially available ultrasound scanner, according to the American Society of Echocardiography (ASE) recommendations for a comprehensive examination.
Diagnostic Test: Echocardiography — As soon as possible following completion of the CPET, subjects will be placed in the supine position and 2D echocardiographic images will be obtained in the apical 4-/ 3-/2-chamber views.

SUMMARY:
The purpose of this study is to find out how much oxygen is used during a cardiopulmonary exercise test (CPET) in women who have mild cardiotoxicity after standard treatment for HER2-positive breast cancer, and to see whether the results of this test can be used to predict how well participants' heart and lungs will work if they continue to receive this kind of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Female
* Diagnosed with a HER2-positive solid tumor (stage I-IV)
* Left ventricular dysfunction prior to the start of HER2-targeted therapy, defined by a LVEF < 53% (or lower limit of normal), or diagnosed with mild cardiotoxicity associated with HER2-targeted therapy, defined by an absolute decrease in LVEF ≥ 10% from pre-treatment to < 53%
* Planning to undergo treatment with HER2-targeted therapy (e.g. trastuzumab, pertuzumab, or ado-trastuzumab) for a minimum of 3 months (i.e. 4 cycles administered every 3 weeks).
* Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Symptomatic heart failure (New York Heart Association Class III or IV)
* Subjects must not have any of the following absolute contraindications to cardiopulmonary exercise testing:

  * Acute myocardial infarction (within 30 days of any planned study procedures),
  * Unstable angina
  * Uncontrolled arrhythmias causing symptoms or hemodynamic compromise,
  * Symptomatic severe aortic stenosis
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Acute pulmonary embolus or pulmonary infarction (within 3 months of any planned study procedures)
  * Thrombosis of lower extremities (within 3 months of any planned study procedures)
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Room air desaturation at rest ≤ 85%
  * Respiratory failure
  * Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
  * Mental impairment leading to inability to cooperate.
* Enrollment onto any other interventional investigational study
* Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research participants will be identified by a member of the participant's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering Cancer Center (MSK). If the investigator is a member of the treatment team, s/he will screen their potential participant's medical records for suitable research study participants and discuss with the subject their potential for enrolling in the research study.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Baseline VO2peak in participants with HER2-positive breast cancer | At baseline
  The primary purpose is to evaluate baseline VO2peak in patients with HER2-positive solid tumors and left ventricular systolic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org